CLINICAL TRIAL: NCT00764582
Title: A Randomized, Observer-masked, Parallel-group, Multicenter Trial Evaluating the Ocular Penetration of 1.5% Levofloxacin Ophthalmic Solution and 0.5% Moxifloxacin Ophthalmic Solution in Subjects Undergoing Corneal Transplant Surgery
Brief Title: Ocular Penetration of 1.5% Levofloxacin and 0.5% Moxifloxacin During Corneal Transplant Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to lack of enrollment.
Sponsor: Santen Inc. (Industry)
Collaborators: Vistakon Pharmaceuticals (Industry)
Responsible Party: Brian Schwam, MD, VISTAKON Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VPH0109
Record Dates: First submitted 2008-09-26; First posted 2008-10-02 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Corneal Transplantation
Keywords: Corneal penetration of levofloxacin and moxifloxacin
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: 1.5% levofloxacin ophthalmic solution
- 2 (Active Comparator)
  Interventions: Drug: 0.5% moxifloxacin ophthalmic solution

INTERVENTIONS:
Drug: 1.5% levofloxacin ophthalmic solution — Topical application Instill 1 drop two times, 5 minutes apart. Time from last drop to surgery is determined by group.
  Group 1: 30 minutes prior to surgery
  Group 2: 1 hour prior to surgery
  Group 3: 2 hours prior to surgery
  Group 4: 4 hours prior to surgery
  Other Names: IQUIX
  Arms: 1
Drug: 0.5% moxifloxacin ophthalmic solution — Topical application Instill 1 drop two times, 5 minutes apart. Time from last drop to surgery is determined by group.
  Group 5: 30 minutes prior to surgery
  Group 6: 1 hour prior to surgery
  Group 7: 2 hours prior to surgery
  Group 8: 4 hours prior to surgery
  Other Names: VIGAMOX
  Arms: 2

SUMMARY:
Compare the corneal penetration of levofloxacin 1.5% and moxifloxacin 0.5% in patients undergoing penetrating keratoplasty (PK)

ELIGIBILITY:
Inclusion Criteria

* Man or woman 18 years of age or older
* Scheduled for corneal transplant surgery
* Patients must be healthy enough to undergo surgery
* Women must be postmenopausal for at least 1 year or surgically sterile incapable of pregnancy
* Women must be abstinent at the discretion of the investigator
* Women practicing an effective method of birth control
* Women agree before entry to continue to use the same method of contraception throughout the study
* Women of childbearing potential must have a negative urine pregnancy test at screening

Exclusion Criteria

* Presence of an active ocular infection or positive history of ocular herpetic infection
* History of severe dry eye syndrome
* Use of contact lenses in the 2 weeks prior to the study and for the duration of the study
* Received an experimental drug or used an experimental medical device within 30 days before the planned start of treatment
* Pregnant or breast feeding
* Employees of the investigator or study center with direct involvement in the proposed study or other studies under the direction of that investigator or study center as well as family members of the employees or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Concentration of levofloxacin and moxifloxacin in the corneal tissue | Time of surgery

SECONDARY OUTCOMES:
Adverse Events | 4 days

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Boynton Beach, Florida
  - Indianapolis, Indiana
  - Great Rapids, Michigan
  - Kansas City, Missouri
  - Springfield, Missouri
  - Stony Brook, New York
  - Cincinnati, Ohio
  - Portland, Oregon